CLINICAL TRIAL: NCT03886545
Title: Objective Assessment for Caregivers With Work-related Musculoskeletal Disorders of the Shoulder
Acronym: AWMSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hopital La Musse (Other)
Responsible Party: Principal Investigator, M. Gilliaux, Principal investigator, Hopital La Musse
Other Study IDs: AWMSD
Record Dates: First submitted 2019-03-19; First posted 2019-03-22 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Musculoskeletal Disorder
Keywords: Assessment ; work-related musculoskeletal disorders of the shoulder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- caregivers with shoulder pain
  Interventions: Other: Assessment of physical and functional capacities
- Healthy subjects
  Interventions: Other: Assessment of physical and functional capacities

INTERVENTIONS:
Other: Assessment of physical and functional capacities — Comparaison of physical and functional capacities between caregivers with work-related musculoskeletal disorders of the shoulder healthy subjects matched in age and gender;

SUMMARY:
Work-related musculoskeletal disorders (WMSD) are a major public health problem both in France and internationally. Our clinical research project focuses on WMSD of the shoulder (WMSD-S), which account for 32% and 23% of these disorders in France and Europe, respectively. In order to prevent WMSD-S, the assessment and rehabilitation of workers' physical and functional capacities (PFC) (e.g. joint amplitude) may complement current interventions (e.g. ergonomics) in a novel manner. As a result, the objectives of this project would be to conduct a cohort study assessing the PFC of caregivers with WMSD-S compared to those of healthy subjects and a randomised, controlled, single-blind, multicentre clinical study assessing the relevance of a rehabilitation program for caregivers with WMSD-S working in a hospital setting. This project would foster the promotion of evidence-based physiotherapy and lead to the development of a interdisciplinary research team dedicated to rehabilitation.

DETAILED DESCRIPTION:
Work-related musculoskeletal disorders (WMSD) are "a set of peri-articular conditions that can affect various structures of the upper limbs, lower limbs and back: tendons, muscles, joints, nerves and the vascular system"(1). WMSD are a major public health problem both in France and internationally. Indeed, these disorders represent 85% of occupational diseases in France (2). Our research project focuses on WMSD-S representing 32% and 23% of these disorders in France (3) and Europe (4), respectively. These shoulder disorders lead to a decrease in the quality of life of workers (2) but also have direct (e.g. 50K € for shoulder tendinitis [ST]) and indirect (e.g. between 100K and 350K € for ST) costs (5).

To prevent WMSD-S, current recommendations encourage regular assessments and interventions at the workers workstation (e.g. biomechanical constraints, ergonomics, etc.) (6,7), their organisation (e. g. "job rotation"...) (8) and psycho-social factors (e. g. stress...) (9) related to work. WMSD-S), which account for 32% and 23% of these disorders in France and Europe, respectively. In order to prevent WMSD-S, the assessment and rehabilitation of workers' physical and functional capacities (PFC) (e.g. joint amplitude) may complement current interventions (e.g. ergonomics) in a novel manner.

It is believed that the assessment of PFC in workers suffering from WMSD-S is essential to better understand the origin of these disorders, and therefore to optimise their care (10) . To our knowledge, no clinical studies have analysed the interest of a protocol for the assessment of WMSD-S in caregivers. From this observation, the first part of this project would consist of a cohort study assessing the PFC of caregivers with WMSD-S, compared to those of healthy subjects matched in age and gender. This study would improve the understanding of the worker's physical and functional impairments; a fundamental aspect for the individualised person-focused interventions (i.e. rehabilitation), in addition to those carried out at the workstation level (i.e. ergonomics).

ELIGIBILITY:
Inclusion Criteria:

* For caregivers with shoulder pain, the inclusion criteria would be: aged between 18 and 65; being a caregiver in a hospital department and having WMSD-S, objectified by shoulder pain.
* For healthy subjects , the inclusion criteria would be : aged between 18 and 65 and no shoulder pain (0/10 on visual analogic scale) in the last 3 months, both at rest and during activity.

Exclusion Criteria:

* For caregivers with shoulder pain, The exclusion criterion would be any traumatic event not related to the professional activity that could impair the functionality of the upper limbs.
* For healthy subject, the exclusion criterion would be any injury to shoulder muscles or tendons.
* For both groups, the exclusion criteria would include smoking, being pregnant, and engaging in traumatic physical activity of the shoulder and any systemic disease or neurological injury.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups
  * experimental group, caregivers with shoulder pain
  * control group, healthy subjects without shoulder pain
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-11-17 (Actual); Primary Completion 2020-11-17 (Actual); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Amplitude | 5 minutes
  shoulder amplitude (in °) computed with inertial sensors
Speed | 5 minutes
  shoulder speed (in °/seconde) computed with inertial sensors
Smoothness | 5 minutes
  shoulder smoothness (peak speed/mean speed) computed with inertial sensors

SECONDARY OUTCOMES:
surface electromyographs | 15 minutes
  fatigability of shoulder muscles assessed using surface electromyographs
global dexterity | 5 minutes
  global manual dexterity quantified using the Box and Block Test
fine manual dexterity | 5 minutes
  fine manual dexterity quantified using Purdue Pegboard Test
activity limitations | 5 minutes
  activity limitations assessed using the "Patient-Specific Functional Scale" questionnaire
participation restrictions | 5 min
  participation restrictions assessed using the "Quick Dash" questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital La Musse, Saint-Sébastien-de-Morsent, France

IPD SHARING:
Plan to Share IPD: No
The data collected will be anonymized, computerized and stored by Maxime GILLIAUX. Only the investigators (Mr GILLIAUX and Mrs Julie VAN NIEUWENHOVE) will have access to the anonymized data in order to carry out the statistical work of this research.

REFERENCES:
- [Background] DGAFP. Guide pratique-Démarche de prévention des troubles musculo-squelettiques.2015; 1-65.
- [Background] DIRECCTE de Normandie. Plan santé au travail 2016-2020 Normandie. oct 2017.
- [Background] INRS. Troubles musculosquelettiques (TMS). INRS; 2015.
- [Background] Schneider et al. OSH in figures: Work-related musculoskeletal disorders in the EU. 2010.
- [Background] ARS Haute-Normandie. Prévenir durablement les Troubles Musculo-Squelettiques. 2013
- [Background] Akkas O, Lee CH, Hu YH, Harris Adamson C, Rempel D, Radwin RG. Measuring exertion time, duty cycle and hand activity level for industrial tasks using computer vision. Ergonomics. 2017 Dec;60(12):1730-1738. doi: 10.1080/00140139.2017.1346208. Epub 2017 Jul 6. PMID 28640656
- [Background] Ghasemi MS, Hosseinzadeh P, Zamani F, Ahmadpoor H, Dehghan N. Ergonomic design and evaluation of a diagnostic ultrasound transducer holder. Int J Occup Saf Ergon. 2017 Dec;23(4):519-523. doi: 10.1080/10803548.2016.1216763. Epub 2016 Sep 7. PMID 27488732
- [Background] Padula RS, Comper MLC, Sparer EH, Dennerlein JT. Job rotation designed to prevent musculoskeletal disorders and control risk in manufacturing industries: A systematic review. Appl Ergon. 2017 Jan;58:386-397. doi: 10.1016/j.apergo.2016.07.018. Epub 2016 Aug 9. PMID 27633235
- [Background] Pransky G, Robertson MM, Moon SD. Stress and work-related upper extremity disorders: implications for prevention and management. Am J Ind Med. 2002 May;41(5):443-55. doi: 10.1002/ajim.10040. PMID 12071496
- [Background] Gutenbrunner C, Meyer T, Melvin J, Stucki G. Towards a conceptual description of Physical and Rehabilitation Medicine. J Rehabil Med. 2011 Sep;43(9):760-4. doi: 10.2340/16501977-0866. PMID 21874211
- [Background] van den Noort JC, Wiertsema SH, Hekman KMC, Schonhuth CP, Dekker J, Harlaar J. Reliability and precision of 3D wireless measurement of scapular kinematics. Med Biol Eng Comput. 2014 Nov;52(11):921-931. doi: 10.1007/s11517-014-1186-2. Epub 2014 Sep 6. PMID 25192921
- [Background] Krause DA, Neuger MD, Lambert KA, Johnson AE, DeVinny HA, Hollman JH. Effects of examiner strength on reliability of hip-strength testing using a handheld dynamometer. J Sport Rehabil. 2014 Feb;23(1):56-64. doi: 10.1123/jsr.2012-0070. Epub 2013 Nov 14. PMID 24231811
- [Background] De Baets L, van der Straaten R, Matheve T, Timmermans A. Shoulder assessment according to the international classification of functioning by means of inertial sensor technologies: A systematic review. Gait Posture. 2017 Sep;57:278-294. doi: 10.1016/j.gaitpost.2017.06.025. Epub 2017 Jun 27. PMID 28683420
- [Background] Seitz AL, Uhl TL. Reliability and minimal detectable change in scapulothoracic neuromuscular activity. J Electromyogr Kinesiol. 2012 Dec;22(6):968-74. doi: 10.1016/j.jelekin.2012.05.003. Epub 2012 Jun 8. PMID 22683057
- [Background] Sivan M, O'Connor RJ, Makower S, Levesley M, Bhakta B. Systematic review of outcome measures used in the evaluation of robot-assisted upper limb exercise in stroke. J Rehabil Med. 2011 Feb;43(3):181-9. doi: 10.2340/16501977-0674. PMID 21305232
- [Background] Hefford C, Abbott JH, Arnold R, Baxter GD. The patient-specific functional scale: validity, reliability, and responsiveness in patients with upper extremity musculoskeletal problems. J Orthop Sports Phys Ther. 2012 Feb;42(2):56-65. doi: 10.2519/jospt.2012.3953. Epub 2012 Feb 1. PMID 22333510
- [Background] Fayad F, Lefevre-Colau MM, Gautheron V, Mace Y, Fermanian J, Mayoux-Benhamou A, Roren A, Rannou F, Roby-Brami A, Revel M, Poiraudeau S. Reliability, validity and responsiveness of the French version of the questionnaire Quick Disability of the Arm, Shoulder and Hand in shoulder disorders. Man Ther. 2009 Apr;14(2):206-12. doi: 10.1016/j.math.2008.01.013. Epub 2008 Apr 23. PMID 18436467